CLINICAL TRIAL: NCT04656834
Title: Hand Surgical Incision Outcomes
Brief Title: Hand Incision Study
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Sponsor
Other Study IDs: AILY20D.947
Record Dates: First submitted 2020-11-23; First posted 2020-12-07 (Actual); Last update posted 2020-12-07 (Actual); Status verified 2020-12

CONDITIONS: Hand Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hand incision closure type 1: The participating surgeon closes the hand surgical incision via the standard method based on personal preference: buried monocryl sutures and skin glue
  Interventions: Procedure: hand incision closure using monocryl sutures and skin glue
- Hand incision closure type 2: The participating surgeon closes the hand surgical incision via the standard method based on personal preference: simple nylon sutures
  Interventions: Procedure: hand incision closure using simple nylon sutures

INTERVENTIONS:
Procedure: hand incision closure using monocryl sutures and skin glue — At the end of surgery, the investigator will close the incision using monocryl sutures and skin glue
  Groups: Hand incision closure type 1
Procedure: hand incision closure using simple nylon sutures — At the end of surgery, the investigator will close the incision using simple nylon sutures
  Groups: Hand incision closure type 2

SUMMARY:
The cosmetic outcome of a patient's surgical scar is important for patient satisfaction, especially in more visibly exposed areas of the body such as the hand. A patient's surgical scar often serves as a long-term reminder of their surgery experience, so optimizing final scar appearance should be of high importance. Surgical incision closure techniques and suture materials may vary by individual hand surgeons, even with common hand procedures.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years old
* Able to provide consent
* Undergoing either trigger finger release or carpal tunnel release

Exclusion Criteria:

* Patients < 18 years old
* Unable to provide consent
* Unable to comply with follow up requirements

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants who are 18 years old or older who are having surgery for either a trigger finger release or carpal tunnel release by one of Rothman Orthopaedics Hand & Wrist Surgeons
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2020-11-30 (Estimated); Primary Completion 2021-11-30 (Estimated); Study Completion 2021-11-30 (Estimated)

PRIMARY OUTCOMES:
Participant Satisfaction with Scar Appearance (Questionnaire #1) | 12 weeks
  Participant will be asked to answer a series of questions regarding the cosmetic appearance of their surgical scar and how satisfied they are with the appearance of the scar as measured by the Patient Scar Assessment Questionnaire (PSAQ).
Participant Satisfaction with Scar Appearance (Questionnaire #2) | 12 weeks
  Participant will be asked to answer a series of questions regarding the cosmetic appearance of their surgical scar and how satisfied they are with the appearance of the scar as measured by the Stony Brook Scar Evaluation Scale (SBSES)
Participant Satisfaction with Scar Appearance (Questionnaire #3) | 12 weeks
  Participant will be asked to answer a series of questions regarding the cosmetic appearance of their surgical scar and how satisfied they are with the appearance of the scar as measured by the Visual Analog Scale (VAS)

CONTACTS AND LOCATIONS:
Locations (1):
- Rothman Orthopaedic Institute, Philadelphia, Pennsylvania, United States